CLINICAL TRIAL: NCT06581289
Title: Cardiac Anesthesia Registry Including Biosignal Database for Prognostication of Postoperative Renal Outcome: Cardiac Anesthesia Renal Outcome in Severance Cardiovascular Hospital - DataBase (CARS-DB)
Brief Title: Cardiac Anesthesia Registry Including Biosignal Database for Prognostication of Postoperative Renal Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0557
Record Dates: First submitted 2024-06-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Anaesthesia
Keywords: Acute Kidney Injury; Cardiovascular Surgical Procedures; Cardiopulmonary Bypass; Biomarker; Biosignal data; Renal outcome
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesia for cardiovascular surgery using cardiopulmonary bypass: patients scheduled for cardiovascular surgery with CPB which requires anesthesia in the operating room

SUMMARY:
AKI(Acute Kidney Injury) is a common complication after cardiac surgery which is associated with increased mortality and morbidity. Collecting perioperative biosignal data and studying their association with renal outcomes can help improve kidney injury, mortality, and morbidity in cardiac surgical patients. Furthermore, the occurrence of AKI, length of hospital stay, and recovery of renal function after discharge are closely associated with the development of chronic kidney disease (CKD). Therefore, regular monitoring of renal function and related indicators in cardiac surgical patients can help improve long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years and older scheduled for cardiac surgery using CPB

Exclusion Criteria:

* emergency operation, the patient is foreigner or illiterate and unable to read the consent form

Ages: 19 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 19 year and older admitted to Severance cardiovascular hospital for cardiac surgery using CPB (Cardiopulmonary bypass).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2034-08-01 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
post-operative AKI incidence within 1 week after cardiac surgery with CPB | within first 7 days after surgery
  The definition of AKI refers to Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury.

SECONDARY OUTCOMES:
MAKE 30 (Major adverse kidney event within 30 days) | within 30 days after surgery
  death, starting dialysis, or decrease in eGFR of 25 % or more within 30 days after surgery
MAKE 90 (Major Adverse kidney event within 90 days) | within 90 days after surgery
  death, starting dialysis, or decrease in eGFR of 25 % or more within 90 days after surgery
incidence of CKD (chronic kidney disease) within 1 year | within 1 year after surgery
  at least one of the following criteria is met, with structural or functional abnormalities of the kidney persisting for at least 3 months within 1 year
  * urine albumin/creatinine ratio ≥ 30 mg/g
  * abnormality in urine sediment test or persistent hematuria
  * renal structural abnormalities found in image study
  * eGFR < 60 ml/min/1.73m2 (GFR category G3a-G5)
1 year mortality | within 1 year after surgery
  death due to any cause within 1 year
in-hospital mortality | from day of hospitalization for surgery until discharge after surgery 1year
  death which occurs during the hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No